CLINICAL TRIAL: NCT04794933
Title: The Effects of Different Proprioceptive Neuromuscular Facilitation Patterns on Pain, Postural Changes and Functionality in Patients With Subacromial Impingement Syndrome: A Randomized Controlled Trial
Brief Title: PNF in Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Ertuğrul Demirdel, Assistant Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Subacromial Impingement Syndrome
Keywords: subacromial impingement; posture; pain; Proprioceptive Neuromuscular Facilitation
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain

STUDY DESIGN:
Intervention Model Description: Patients who met the inclusion criteria and agreed to participate were randomly allocated to Group 1 [Conventional therapy (CT)], Group 2 [CT+ PNF in extremity pattern] and Group 3 [CT+ PNF in extremity pattern+PNF in scapula and upper trunk patterns].
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional therapy (CT) (Active Comparator): Cold pack (15 minutes); pulsed ultrasound therapy (1 watt/cm², 3 MHz, 1:2 pulsed mode; 3 minutes); transcutaneous electrical nerve stimulation (60-120 Hz; 20 minutes) and exercises (20 minutes). The exercises included stretching, strengthening and posture exercises.
  Interventions: Other: Conventional therapy
- CT+ PNF in extremity pattern (Experimental): PNF in the extremity pattern, were instructed to actively move through the PNF flexion-abduction-external rotation diagonal pattern for 10 repetitions with manual facilitation and the treatment was performed within the range in which pain did not occur. Rhythmic stabilization and repeated contractions were applied from the PNF techniques.
  Interventions: Other: Conventional therapy; Other: CT+ PNF in extremity pattern
- CT+ PNF in extremity pattern+PNF in scapula and upper trunk patterns (Experimental): PNF in scapula and upper trunk patterns in addition to PNF in the extremity pattern. The scapular pattern application was performed by positioning the affected extremity in a relaxed position above the stable side in the side-lying position. Rhythmic stabilization and repeated contractions were applied from the anterior-elevation position in the direction of posterior-depression. Extension, lateral flexion and rotation to the affected side were performed in the trunk patterns in rhythmic stabilization and repeated contractions.
  Interventions: Other: Conventional therapy; Other: CT+ PNF in extremity pattern; Other: CT+ PNF in extremity pattern+PNF in scapula and upper trunk patterns

INTERVENTIONS:
Other: Conventional therapy
Other: CT+ PNF in extremity pattern
  Arms: CT+ PNF in extremity pattern; CT+ PNF in extremity pattern+PNF in scapula and upper trunk patterns
Other: CT+ PNF in extremity pattern+PNF in scapula and upper trunk patterns
  Arms: CT+ PNF in extremity pattern+PNF in scapula and upper trunk patterns

SUMMARY:
Although proprioceptive neuromuscular facilitation (PNF) techniques have been used in the treatment of different shoulder problems, PNF techniques in scapular and upper trunk patterns with extremity pattern have not been considered as a possible option for the treatment of Subacromial Impingement Syndrome (SIS). The aim of this study was to evaluate the effects of different PNF patterns in SIS.

DETAILED DESCRIPTION:
This randomized controlled trial was conducted in the Outpatient Clinic of a Physiotherapy and Rehabilitation Department in Ankara, Turkey. The demographic and clinical characteristics of the patients were recorded. Voluntary patients with SIS were regarded as eligible for the study if they met the inclusion criteria. Pain, posture and functionality were assessed before and after intervention. Patients who met the inclusion criteria and agreed to participate were randomly allocated to Group 1 [Conventional therapy (CT)], Group 2 [CT+ PNF in extremity pattern] and Group 3 [CT+ PNF in extremity pattern+PNF in scapula and upper trunk patterns]. A simple randomization method was used with opaque sealed envelopes containing "A", "B" or "C". Group allocation was performed by an independent therapist, not involved in the study. All patients received physiotherapy for approximately 60 mins each session, 3 sessions per week for 6 weeks. Conventional therapy consisted of cold pack (15 minutes); pulsed ultrasound therapy (1 watt/cm², 3 MHz, 1:2 pulsed mode; 3 minutes); transcutaneous electrical nerve stimulation (60-120 Hz; 20 minutes) and exercises (20 minutes). The exercises included stretching, strengthening and posture exercises. The exercises, and the duration and intensity of conventional physiotherapy were selected according to previous studies which showed that a physiotherapy program 3 times a week for 6 weeks was effective in improving function and relieving pain in SIS. The physiotherapy program was applied to all patients at the same intensity by the same physiotherapist and patients did the exercises every day throughout the 6-week period. The patients were also advised to avoid overhead activities.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with SIS,
* aged between 18 and 65 years,
* shoulder pain ongoing for more than four weeks,
* loss of active shoulder motion or painful ROM,
* no treatment related to the shoulder in the last 6 months.

Exclusion Criteria:

* history of frozen shoulder,
* disorders of the acromioclavicular joint,
* possession of a curved or hooked acromion,
* shoulder instability,
* degenerative arthritis of the glenohumeral joint,
* calcifying tendonitis,
* post-traumatic disorders,
* shoulder surgery and/or elbow, hand, wrist and cervical spine disorders,
* diseases that can cause positional vertigo.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Scapular stability | Change from baseline scapular stability at 6 weeks
  The lateral scapular slide test (LSST) was applied to evaluate scapular stability. In the first position (LSST 1), both arms are relaxed at the sides with the glenohumeral joint in a neutral position. In the second position (LSST 2), the subject places both hands on the ipsilateral hips with the humerus in medial rotation in 45° of abduction in the coronal plane. In position 3 (LSST 3), the subject actively extends both elbows and places the upper extremities in a position of maximum medial rotation in 90° of abduction in the coronal plane. The inferomedial angle of the scapula is palpated and marked on both the affected and unaffected sides, and the spinous process of the thoracic vertebra in the same horizontal plane (the reference vertebra) is then marked. The measurements from the reference point on the spine to the medial border of the scapula are measured on both sides in all 3 test positions.
Anterior tilt of the head | Change from baseline anterior tilt of the head at 6 weeks
  The distance was measured from the sternal notch to the tip of the chin with a tape measure.
Rounded shoulder | Change from baseline rounded shoulder at 6 weeks
  The subject stood in a relaxed position with their heels against a wall. The posterolateral acromion was marked and the ruler was held square. The measurement was taken from the acromion to the wall behind the subject to determine the amount of forward displacement.
Thoracic kyphosis | Change from baseline thoracic kyphosis at 6 weeks
  The gravity-dependent inclinometer (BASELINEᴿ Bubble inclinometer-USA) was used to measure kyphosis. In the first measurement, the inclinometer was placed over the region of the 1st and 2nd thoracic spinous processes and in the second, over the region of the 12th thoracic and 1st lumbar spinous processes. The total of the angles in each measurement was recorded.

SECONDARY OUTCOMES:
Pain severity | Just before the treatment and at the end of 6-week treatment
  Patients' pain will be assessed for three different situations: "at rest", "at activity" and "at night" before and after treatment. The patient is asked to mark the severity of pain on the 10 cm horizontal line [left end(0) = no pain, right end(10)= unbearable pain ]. Data is measured with a standard ruler and results are recorded in centimeters (cm).
Functional status | Just before the treatment and at the end of 6-week treatment
  The numerically-scaled Shoulder Pain and Disability Index, a 13-item self-administered instrument measuring shoulder functional status, was used.

CONTACTS AND LOCATIONS:
Overall Officials: Ertuğrul Demirdel, PhD, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cools AM, Struyf F, De Mey K, Maenhout A, Castelein B, Cagnie B. Rehabilitation of scapular dyskinesis: from the office worker to the elite overhead athlete. Br J Sports Med. 2014 Apr;48(8):692-7. doi: 10.1136/bjsports-2013-092148. Epub 2013 May 18. PMID 23687006
- [Background] Escamilla RF, Yamashiro K, Paulos L, Andrews JR. Shoulder muscle activity and function in common shoulder rehabilitation exercises. Sports Med. 2009;39(8):663-85. doi: 10.2165/00007256-200939080-00004. PMID 19769415
- [Background] Green S, Buchbinder R, Hetrick S. Physiotherapy interventions for shoulder pain. Cochrane Database Syst Rev. 2003;2003(2):CD004258. doi: 10.1002/14651858.CD004258. PMID 12804509
- [Background] Gumina S, Di Giorgio G, Postacchini F, Postacchini R. Subacromial space in adult patients with thoracic hyperkyphosis and in healthy volunteers. Chir Organi Mov. 2008 Feb;91(2):93-6. doi: 10.1007/s12306-007-0016-1. Epub 2008 Mar 3. PMID 18320381
- [Background] Hanratty CE, McVeigh JG, Kerr DP, Basford JR, Finch MB, Pendleton A, Sim J. The effectiveness of physiotherapy exercises in subacromial impingement syndrome: a systematic review and meta-analysis. Semin Arthritis Rheum. 2012 Dec;42(3):297-316. doi: 10.1016/j.semarthrit.2012.03.015. Epub 2012 May 18. PMID 22607807
- [Background] Hickey D, Solvig V, Cavalheri V, Harrold M, Mckenna L. Scapular dyskinesis increases the risk of future shoulder pain by 43% in asymptomatic athletes: a systematic review and meta-analysis. Br J Sports Med. 2018 Jan;52(2):102-110. doi: 10.1136/bjsports-2017-097559. Epub 2017 Jul 22. PMID 28735288
- [Background] Holmgren T, Hallgren HB, Oberg B, Adolfsson L, Johansson K. Effect of specific exercise strategy on need for surgery in patients with subacromial impingement syndrome: randomised controlled study. Br J Sports Med. 2014 Oct;48(19):1456-7. doi: 10.1136/bjsports-2014-e787rep. PMID 25213604
- [Background] Hunter DJ, Rivett DA, McKeirnan S, Smith L, Snodgrass SJ. Relationship Between Shoulder Impingement Syndrome and Thoracic Posture. Phys Ther. 2020 Apr 17;100(4):677-686. doi: 10.1093/ptj/pzz182. PMID 31825488